CLINICAL TRIAL: NCT07288437
Title: Adaptive Deep Brain Stimulation Targeting the Dentate Nucleus to Treat Spinocerebellar Ataxia
Brief Title: Deep Brain Stimulation for Spinocerebellar Ataxia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Raynor Cerebellum Project (Unknown)
Responsible Party: Principal Investigator, Marta San Luciano Palenzuela, MD, Professor of Neurology, University of California, San Francisco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-44582
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Spinocerebellar Ataxia (SCA); Spinocerebellar Ataxia Type 6
Keywords: adaptive deep brain stimulation; aDBS; Spinocerebellar Ataxia; Spinocerebellar Ataxia Type 6; SCA6; DBS; deep brain stimulation
MeSH Terms: conditions — Spinocerebellar Ataxias | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Adaptive Deep Brain Stimulation (aDBS) (Experimental): One month after patients undergo DBS surgery in the cerebellum, conventional deep brain stimulation (cDBS) programming will begin to identify stimulation parameters (such as amplitude, contact, frequency, and pulse width) and ensure no adverse wide effects are witness. This phase also allows the study team to make sure device and electrode placement are working as intended. About nine months after implantation, the investigators will switch system settings over to aDBS to evaluate the feasibility, safety, and tolerability in the dentate nucleus of the cerebellum. Symptoms and side effects will be assessed by patients' self-reports, validated clinical scales, and wearable devices, which will be used to track movements and sleep data.
  Interventions: Device: Deep Brain Stimulation (DBS)

INTERVENTIONS:
Device: Deep Brain Stimulation (DBS) — This device will be surgically implanted into the dentate nucleus of the cerebellum.
  Other Names: Medtronic Percept

SUMMARY:
The goal of this clinical trial is to test the safety of placing Deep Brain Stimulators (DBS) in the cerebellum and using electrical stimulation of that part of the brain to treat symptoms related to the participants spinocerebellar ataxia. Five adults diagnosed with spinocerebellar ataxia type 6 (SCA6) with inadequate cerebellar symptom relief will be implanted with a Medtronic Percept Primary Cell Neurostimulator. The device will be implanted into the dentate nucleus, which is a structure located within the cerebellum that is responsible for controlling movement and balance.

Specifically, the investigators will be using adaptive deep brain stimulation (aDBS), which analyzes brain signals and automatically adjusts the strength, timing, and pattern of stimulation according to the patient's needs at any given moment. This study will evaluate the feasibility, safety, and tolerability of aDBS in SCA6 patients.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of SCA6 by a Movement Disorders specialist following established criteria recommended by the Movement Disorders Society.
2. A positive genetic test for SCA6.
3. A total scale ≥ 8 on the Scale of the Assessment and Rating of Ataxia (SARA) rating scale.
4. Ability to walk with or without support (score < 8 on the 'gait' subsection of the SARA rating scale).
5. Age ≥ 21 years and < 89 years.
6. Ability to give informed consent for the study.
7. Be able to understand the study protocol.

Exclusion Criteria:

1. Inability or unwillingness to comply with the study protocol.
2. History of previously implanted neurostimulators, pacemakers, defibrillators, or metallic head implants.
3. Severe cognitive impairment or dementia, defined as a score < 21 on the Montreal Cognitive Assessment (MoCA).
4. Evidence of ataxia due to other etiologies, including but not limited to:

   1. Genetic/inherited disorders other than SCA6.
   2. Acquired causes: tramautic brain injury, multiple sclerosis, paraneplastic cerebellar degeneration, infections or post-infectious cerebellitis, autoimmune ataxias (e.g., anti-GAD, gluten ataxia).
   3. Toxic/metabolic causes: alcoholic cerebellar degeneration, vitamin deficiencies.
   4. Structural, vascular, or neoplastic causes: cerebellar stroke, tumors, congenital malformations.
   5. Suspected multiple system atrophy-cerebellar type (MSA-C).
5. The presence of active and untreated psychiatric illness, severe depression (Beck Depression Inventory ≥ 21), or personality disorder at the discretion of the study team.
6. Coagulopathy, uncontrolled epilepsy, or other medical condition considered to place the patient at elevated risk for surgical complications. Presence of a concomitant medical condition that, in the investigator's opinion, may interfere with the study participation or gait/balance, for example, severe arthritis.
7. Presence of a concominant medical condition that, in the investigator's opinion, may interfere with the study participation or gait/balance, for example, severe arthritis.
8. Requirement of diathermy, electroconvulsive therapy, or transcranial magnetic stimulation.
9. Pregnancy or lactation.
10. Active suicidal ideation, defined as fined as a "Yes" response to questions #2-5 on the Columbia Suicide Severity Rating Scale, C-SSRS.
11. Refractory Epilepsy.

Ages: 21 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2029-03 (Estimated); Study Completion 2031-03 (Estimated)

PRIMARY OUTCOMES:
Average total score for the Assessment and Rating of Ataxia (SARA) | From baseline through study completion, about 2 years.
  SARA is a clinical scale that assesses a variety of different impairments for individuals with cerebellar ataxia. The scale includes 8 different items that are related to gait, stance, sitting, speech, finger-chase test, nose-finger test, fast alternating movements, and heel-shin test. The total amount of points on SARA ranges from 0 (no ataxia) to 40 (most severe ataxia). This study requires participants to have a minimum SARA score of at least 8 so that people who are relatively early in their disease course with limited cerebellar degeneration can be included.
Average total Patient-Reported Outcome Measure of Ataxia (PROM-Ataxia) Score | From baseline through study completion, about 2 years.
  PROM-Ataxia is a 3-domain, 70-item questionnaire used for the assessment of ataxia-related symptoms. It incorporates a series of questions ranging to the impact of cerebellar dysfunction on physical abilities, activities of daily living, and cognitive-emotional challenges. The maximum severity score on PROM-Ataxia is 280, where all 70 questions are scored on a 0-4 Likert scale. 0 represents never and 4 represents always.

CONTACTS AND LOCATIONS:
Overall Officials: Marta San Luciano Palenzuela, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No